CLINICAL TRIAL: NCT07279584
Title: An Open-Label, Single-Arm Study to Evaluate the Safety and Efficacy of Golidocitinib Combined With GemOx in the Treatment of Relapsed or Refractory Peripheral T-Cell Lymphoma
Brief Title: Golidocitinib Combined With GemOx in RR PTCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor and Director，Shanghai Institute of Hematology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Golidocitinib Combined
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Peripheral T-cell Lymphomas (PTCL)
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Golidocitinib Combined with GemOx (Experimental)
  Interventions: Drug: golidocitinib; Drug: GEMOX

INTERVENTIONS:
Drug: golidocitinib — 150mg qd po
Drug: GEMOX — Gemcitabine: 1000mg/m2, d1; Oxaliplatin:100mg/m2, d1

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of golidocitinib in combination with the GemOx regimen in r/r PTCL

ELIGIBILITY:
Inclusion Criteria:

1. fully understood and voluntarily signed the ICF for this study
2. aged ≥ 18 years;
3. patients with R/R PTCL who have received at least one prior systemic therapy.
4. Patients must have at least one measurable lesion by computed tomography (CT)/magnetic resonance imaging (MRI) (longest diameter of lymph node lesions > 1.5 cm or longest diameter of extranodal lesions > 1 cm); evaluable lesions: PET-CT examination showed increased local uptake in lymph nodes or extranodal sites (higher than liver) and imaging characteristics consistent with lymphoma performance
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2;
6. Adequate bone marrow function, renal function, liver function: ANC ≥ 1.0 × 109/L, hemoglobin ≥ 8.0 g/dL, platelets ≥ 75 × 109/L Note: if the investigator believes that the patient 's above test values are below the lower limit of the protocol due to lymphoma invading the bone marrow, the patient can be enrolled after assessment.Creatinine clearance > 40 mL/min, calculated by Cockcroft-Gault method: • serum total bilirubin ≤ 1.5 x upper limit of normal (ULN), except for unconjugated bilirubinemia in Gilbert 's syndrome; • ALP (in the absence of bone disease), ALT, and AST ≤ 3.0 × ULN (in the presence of liver metastases, ≤ 5 × ULN); • international normalized ratio (INR) ≤ 1.5 × ULN, or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
7. Current negative for human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or cytomegalovirus (CMV), and inactive if positive:

   * HBV infected patients with positive hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb)] but negative results of HBV DNA polymerase chain reaction (PCR) test can be enrolled; these patients require continuous antiviral therapy after enrollment and HBV DNA PCR test is performed every cycle;
   * Patients with positive HCV serology but negative HCV RNA test may be enrolled;
   * CMV IgM antibody positive,However, patients who tested negative for CMV DNA could be enrolled;
8. female patients of childbearing potential had to agree to use a double contraception method at least 28 days before starting study drug, during treatment, and for 6 months after the last dose of study drug, and male patients with partners of childbearing potential had to also use an effective double contraception method during the study and for 3 months after the last dose of study drug, e.g., condom, sponge plug, foam, contraceptive jelly, diaphragm cap or intrauterine contraceptive device, contraceptive pills (oral or parenteral), contraceptive implant (Implanon ®), injectable intravascular injection, or other contraceptive measures.Postmenopausal women (> 45 years of age and amenorrheic for > 1 year) and surgically sterile women are exempt from this criterion.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria must be excluded from this study:

1. previously used drugs in the treatment regimen may affect the efficacy evaluation of this study (assessed by the investigator)
2. previous bone marrow malignancies, including MDS, AML, MPN, etc.
3. and have clinically significant abnormal test results as judged by the investigator;
4. inability to be orally administered, previous surgical history or severe gastrointestinal diseases such as dysphagia, active gastric ulcer, etc., which the investigator believes may affect the absorption of the study drug;
5. major surgery within 4 weeks before the first study drug administration (referring to grade 3 and 4 surgery as specified in the Measures for the Administration of Clinical Application of Medical Technology implemented on May 1, 2009);
6. current clinically significant active cardiovascular disease, such as uncontrolled arrhythmia, congestive heart failure, any grade 3 or 4 heart disease defined by the New York Heart Association functional classification, or a history of myocardial infarction within 6 months after screening.Left ventricular ejection fraction < 50% measured by echocardiography
7. Venous thrombosis or pulmonary embolism within 3 months before study drug administration;
8. History of stroke or intracranial hemorrhage within 6 months before the first study drug administration;
9. Active infection requiring systemic treatment;
10. History of inflammatory bowel disease (eg, Crohn 's disease or ulcerative colitis);
11. Known hypersensitivity to study drug;
12. Any other disease, metabolic abnormality, physical examination abnormality, or laboratory abnormality of significant clinical significance that, in the judgment of the investigator, gives reason to suspect that the patient has a disease or condition that would make the use of the study drug inappropriate or would compromise the interpretation of the study results or put the patient at high risk.
13. pregnant (positive pregnancy test) or lactating women;
14. patients who have had previous organ transplantation;
15. diagnosed or treated for malignancies other than PTCL, with the following exceptions: a) malignancies treated with curative therapy ≥ 3 years before randomization and without known active disease; b) adequately treated non-melanoma skin cancer or malignancies without evidence of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | Tumor evaluation was assessed at screening and at the end of treatment (around 3 cycles) then every 12-24 weeks until disease progression (each cycle is 21 days) through study completion, an average of 1 year.
  Percentage of participants with complete response partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Progression-free survival | Baseline up to data cut-off(up to approximately 2 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Complete Response Rate | Tumor evaluation was assessed at screening and at the end of treatment (around 3 cycles) then every 12-24 weeks until disease progression (each cycle is 21 days) through study completion, an average of 1 year.
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Duration of Response | Baseline up to data cut-off(up to approximately 2 years)
  Applicable to complete or partial response participants. DoR was defined as the time from the first documented date of complete or partial response until the date of the disease progression or death from any causes.
Overall survival | Baseline up to data cut-off(up to approximately 2 years)
  Percentage of participants with complete or partial response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Adverse Events | Baseline up to data cut-off(up to approximately 3 years)
  Adverse Events are assessed based on CTCAE v5.0

IPD SHARING:
Plan to Share IPD: No